CLINICAL TRIAL: NCT01320423
Title: Surgical Trial in Lobar Intracerebral Haemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Ta Chiu, Graduate Institute of Injury Prevention and Control, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99073
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Intracerebral Haemorrhage
Keywords: Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery (Other)
  Interventions: Procedure: Surgical Trial

INTERVENTIONS:
Procedure: Surgical Trial — Surgical Trial in Lobar Intracerebral Haemorrhage

SUMMARY:
To establish whether a policy of earlier surgical evacuation of the haematoma in selected patients with spontaneous lobar ICH will improve outcome compared to a policy of initial conservative treatment. The trial will also help to better define the indications for early surgery.

This will overcome two of the criticisms of STICH (timing was too late and sometimes location was too deep). The subgroup identified in STICH is clinically sensible and the hypothesis identified for STICH II is in line with current neurosurgical opinion.

DETAILED DESCRIPTION:
STICH II is an international multicentre randomised parallel group trial comparing early craniotomy to evacuate the haematoma with initial conservative treatment, following spontaneous superficial intracerebral haemorrhage affecting the lobar region only. Only patients for whom the treating neurosurgeon is in equipoise about the benefits of early craniotomy compared to initial conservative treatment are eligible for the trial. Outcome is measured at six months via a postal questionnaire including the Glasgow Outcome scale, Modified Rankin Scale, EuroQol and Barthel. Six hundred patients will be recruited to the trial over thirty months. Follow-up will take six months with analysis and reporting taking one year.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a spontaneous lobar ICH on CT scan (1 cm or less from the cortex surface of the brain)
* Patient within 48 hours of ictus
* Best MOTOR score on the GCS of 5 or 6 and best EYE score on the GCS of 2 or more.
* Volume of haematoma between 10 and 100ml [Calculated using (a x b x c)/2 method]

Exclusion Criteria:

* Clear evidence that the haemorrhage is due to an aneurysm or angiographically proven arteriovenous malformation.
* Intraventricular haemorrhage of any sort
* ICH secondary to tumour or trauma.
* Basal ganglia, thalamic, cerebellar or brainstem haemorrhage or extension of a lobar haemorrhage into any of these regions.
* Severe pre-existing physical or mental disability or severe co-morbidity which might interfere with assessment of outcome.
* If surgery cannot be performed within 12 hours.
* If the haematological effects of any previous anticoagulants are not completely reversed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-04 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale/ Modified Rankin Scale | six months
  Unfavourable outcome will be death or severe disability which will be defined using a prognosis based 8 point Glasgow Outcome Scale/ Modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ta Chiu, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan